CLINICAL TRIAL: NCT01507454
Title: Vagifem® Used for the Treatment of Atrophic Vaginitis Due to Oestrogen Deficiency
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: VAG-1935
Record Dates: First submitted 2012-01-05; First posted 2012-01-11 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Menopause; Postmenopausal Vaginal Atrophy
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Local treatment
  Interventions: Drug: estradiol, 25 mcg

INTERVENTIONS:
Drug: estradiol, 25 mcg — Vaginal tablets for 6-12 weeks according to product labelling

SUMMARY:
This study is conducted in Europe. The aim of this study is to investigate the self-reported impact of Vagifem® (estradiol) treatment on urogenital discomfort in women with atrophic vaginitis due to oestrogen deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Atrophic vaginitis due to estrogen deficiency
* Post-menopausal

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with atrophic vaginitis caused by estrogen deficiency prescribed with Vagifem® by their treating physician
Sampling Method: Probability Sample
Enrollment: 1613 (Actual)
Dates: Start 2006-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects reporting vaginal symptoms occuring 'often' and 'frequently'
Percentage of subjects reporting 'moderate' and 'severe' vaginal symptoms

SECONDARY OUTCOMES:
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Mainz, Germany

REFERENCES:
- [Result] Stute P. Urogenitale Beschwerden und Östradioltherapie: Auswirkung einer vaginalen niedrig dosierten Östradioltherapie auf die Prävalenz und Intensität von urogenitalen Beschwerden. Gynäkologische Endokrinologie 2008; 6 (1): 48-52
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com